CLINICAL TRIAL: NCT02968186
Title: Implementing Screening and Brief Interventions for Excessive Drinkers in Primary Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agrupamento de Centros de Saúde de Dão Lafões (Other)
Collaborators: University of Cambridge (Other); University of Stirling (Other); Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Frederico Rosário, Dr., Agrupamento de Centros de Saúde de Dão Lafões
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ASBI-2017
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Alcohol-Related Disorders
Keywords: Mass Screening; Counseling; Primary Health Care
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implementation program (Experimental): Health professionals will receive a training and support implementation program
  Interventions: Behavioral: Implementation program
- Waiting list (No Intervention): Health professionals will be assigned to a waiting list to receive the implementation program

INTERVENTIONS:
Behavioral: Implementation program — Health professionals in the intervention arm will receive up to four training sessions in the first three months of the implementation period. Practice support will be continuously available throughout the project. Posters specifically designed for this project will be added to the primary health care units aiming to facilitate eliciting alcohol issues during the consultations, and to help professionals remembering to conduct alcohol screening and brief intervention. Leaflets to be handed-in to patients were also specifically produced for this project, aiming to aid professionals in advising at-risk drinkers to cut down. The research team will schedule with each primary health care unit regular visits for feedback on the progress of the program.
  Arms: Implementation program

SUMMARY:
The objective of this study is to investigate the efficacy of an implementation program specifically designed to increase alcohol screening and brief intervention rates in primary health care.

DETAILED DESCRIPTION:
Alcohol is an important risk factor for several diseases, even when consumed moderately. Screening and advising at-risk drinkers to cut-down is a highly effective and cost-effective intervention when conducted in primary healthcare settings. However, these interventions are seldom implemented at the primary care level.

Twelve out of the 26 primary health care units of the Dão Lafões Grouping of Primary Health Care Centres will be randomized to two groups: the intervention arm will receive the new implementation program; the control group will be on a waiting list for receiving the implementation program and will receive the intervention after the testing phase of the trial is completed. The study will last for one year, starting in January 2017. The implementation program was designed in order to overcome known barriers for implementing alcohol screening and brief advice in primary health care. The Behaviour Change Wheel and the Theoretical Domains Framework were used to pinpoint the constructs and behaviour change techniques most suited to address the barriers in order to achieve practice changes.

ELIGIBILITY:
Inclusion Criteria:

* Primary health care units of the Dão Lafões Grouping of Primary Health Care Centres (family physicians/general practitioners, family medicine residents, practice nurses and receptionists)

Exclusion Criteria:

* Primary health care units with four or less general practitioners
* Primary health care units that have a specific alcohol program already implemented

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Alcohol screening rate | 12 months
  Percentage of eligible patients visiting the primary health care centre for an appointment with a general practitioner or nurse who were screened for alcohol use with the Alcohol Use Disorders Identification Test

SECONDARY OUTCOMES:
Improvement of general practitioners attitudes toward at-risk drinkers | 12 months
  Short Alcohol and Alcohol Problems Perception Questionnaire given before and after intervention. General practitioners are classified into a more positive or more negative attitudes group based on the answers given. The groups will be compared before and after.
Improvement in knowledge related to alcohol screening and brief intervention | 12 months
  Four multiple choice questions. These questions will measure the theoretical knowledge of health professionals to key concepts related to alcohol screening and brief intervention. The groups will be compared before and after.
Improvement in barriers for implementing alcohol screening and brief intervention | 12 months
  Level of agreement with 33 statements. Each statement can be mapped to a specific domain of the Theoretical Domains Framework. The groups will be compared before and after.
Utility of materials used in the trial | Through study completion, an average of 12 months
  Level of agreement with 6 statements. Participants (intervention arm only) will be asked to rate the impact of the materials that were specifically produced to be used during the trial.
Brief intervention rate | 12 months
  Percentage of patients who screened positive that were offered at least one brief intervention

CONTACTS AND LOCATIONS:
Overall Officials: Frederico M Rosário, MD, Principal Investigator — Dão Lafões Grouping of Primary Health Care Centres
Locations (1):
- Dão Lafões Grouping of Primary Health Care Centres, Viseu, Dão Lafões, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosario F, Vasiljevic M, Pas L, Fitzgerald N, Ribeiro C. Implementing alcohol screening and brief interventions in primary health care: study protocol for a pilot cluster randomized controlled trial. Fam Pract. 2019 Mar 20;36(2):199-205. doi: 10.1093/fampra/cmy062. PMID 29939239